CLINICAL TRIAL: NCT06196554
Title: Exploratory Study of Gastric Cancer Organoids in the Screening of Neoadjuvant Chemotherapy and Immunotherapy Drugs
Brief Title: Gastric Cancer Organoids in the Screening of Neoadjuvant Drugs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Dong Bing Zhao (Other)
Responsible Party: Sponsor-Investigator, Dong Bing Zhao, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Organization: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Other Study IDs: Cancer Institute and Hospital,
Record Dates: First submitted 2023-12-01; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Gastric Cancer; Organoid; Neoadjuvant Therapy
MeSH Terms: conditions — Stomach Neoplasms | interventions — Oxaliplatin; Irinotecan; Fluorouracil; Paclitaxel; pembrolizumab; Nivolumab

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Crushed ice was put into the special box for sampling, and several tissue protection media were prepared and placed in the ice box. The tissues were stored in the sample protection media immediately after isolation and transported to the laboratory. Ice PBS was poured into an ordinary petri dish, and the newly obtained gastric cancer tissue of enrolled patients was removed and cleaned in the dish with long tweezers (if the tissue was large, it could be cut into small pieces for easy cleaning) until clean.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: Oxaliplatin — According to the first-line drugs provided by the NCCN guidelines, the concentration of each drug was added to the organoid culture medium after setting 5-6 concentration gradients according to literature reports. Chemo-sensitive and drug-resistant.
  Construction of gastric cancer organoid T cell co-culture system to screen sensitive immunotherapy drugs.
  Other Names: Irinotecan (SN-38); 5-Fluorouracil; Paclitaxel; Pembrolizumab; Nivolumab

SUMMARY:
Gastric cancer is an important disease burden that threatens human health. Due to the complex biological characteristics of gastric cancer, the research on gastric cancer is still at a low level. Organoid technology is a breakthrough technology in cancer research. Gastric cancer organoid is a good model for gastric cancer research by three-dimensional culture of tumor cells in vitro, which simulates the spatial morphology and structure of tumors in vivo while preserving the biological characteristics of tumor cells. At present, gastric cancer organoid models have shown great advantages in many fields, such as the mechanism of gastric cancer development, tumor drug resistance, large-throughput chemotherapy drug screening, novel therapeutic target searching, and preclinical validation of novel drugs.

In the current clinical trial, investigators cultured organoids from gastroscopic biopsy tissue of gastric cancer patients, and compared the organoids with the sampled tumors, including immunohistochemical indicators (Ki67+/CK20+/CDX2+), WES sequencing results. At the same time according to the guidelines. The recommended treatment plan is to compare the organoid model drug screening results with the clinical drug sensitivity.

DETAILED DESCRIPTION:
There is an important clinical problem in neoadjuvant chemotherapy, adjuvant chemotherapy and palliative chemotherapy for locally advanced gastric cancer, that is, insufficient effectiveness of chemotherapy. Among the patients with neoadjuvant therapy, some patients will have pathological complete remission, and the prognosis of these patients is better than that of other patients.

However, not all patients have a good pathological response after neoadjuvant chemotherapy, although many studies have reported uneven response rates and individual differences in patient sensitivity to chemotherapy drugs. At present, investigators still lack adequate methods to predict the effectiveness of chemotherapy and adjust treatment strategies in time to achieve the best clinical outcomes.

In addition, targeted therapy and immunotherapy are widely used in clinical practice, and gene sequencing is performed on tumor samples of patients to guide the selection of targeted drugs. However, according to clinical data feedback, this method has many limitations, for example, patients with a targeted gene mutation of a targeted drug cannot respond to the drug, while patients without the targeted gene mutation can respond very well to the drug. The reason is that the sequencing results based on some known proto-oncogenes or tumor suppressor genes cannot fully reflect the genomic background of the patient, including some unknown cancer-related genes, and even non-coding protein sequences play important regulatory roles in the process of cancer. Therefore, how to quickly select the most effective drug for this patient among the numerous cancer targeted drugs on the market is the decisive factor for the success or failure of cancer precision medicine.

In recent years, an important breakthrough in basic tumor research is the tumor organoid technology established in vitro, which directly obtains tumor tissue from patients, rapidly expands in vitro, and forms organoids with a high physiological and pathological state similar to the original tissue in a short time. This organoid is a three-dimensional assembly of cells containing more than one cell type. Since the cultured organoids are derived from the patient's own tumor tissue, they can well retain various characteristics of the tumor tissue in situ. Compared with the traditional 2D cell line culture, organoids are directly derived from patients, can retain the patient's genomic information and epigenetic information, maintain the heterogeneous components of the original tumor, and have a 3D structure that is more in line with the conditions in vivo, so it is more representative. Compared with the animal transplant tumor model derived from patients, organoids have the advantages of low cost, high success rate, short culture cycle and easy operation. In general, tumor organoids combine the advantages of 2D cell line culture and animal transplant tumor models, which can not only fully reflect the genetic information and tumor phenotype of patients, but also ensure the heterogeneity of tumors, and have high economic benefits. Therefore, they are favored in scientific research and clinical practice, and are effective tools for evaluating drug response and screening drugs. There are already some of the top cancer research institutes in the world, National Cancer Institute (Netherlands), Cancer Research UK (UK) and the Wellcome Trust Sanger Institute (UK) are working together to build a sample bank of various Tumor organoids that are already being used in precision medicine for cancer patients.

As such, investigators designed a single-center prospective, observational clinical trial for patients with locally advanced gastric cancer, aiming to explore the application of gastric cancer organoids in chemotherapy drug screening, so as to improve the efficacy of neoadjuvant chemotherapy for gastric cancer and provide a basis for the precision treatment of neoadjuvant therapy for gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* 1: The patients voluntarily participated in this study and signed the informed consent;
* 2: 18 to 80 years old.
* 3: American Society of Anesthesiologists (ASA) score ≤3 (no risk of anesthesia during surgery).
* 4: Patients diagnosed with gastric cancer by pathological examination.
* 5: Expected survival is greater than 6 months.
* 6: Blood routine: Hb≥70g/L, WBC≥3.5×109/L, ANC≥1.5×109/L, PLT≥80×109/L.
* 7: Serum ALT and AST≤2×ULN; Serum creatinine≤1.5×ULN.
* 8: Women of childbearing age must undergo a pregnancy test (serum or urine) within 7 days before enrollment, and the result is negative, and they are willing to use appropriate methods of contraception during the trial.
* 9: According to the judgment of the investigator, patients who can comply with the protocol.
* 10: Patients with locally advanced gastric cancer requiring neoadjuvant therapy.

Exclusion Criteria:

* 1: Active or uncontrolled serious infection.
* 2: Liver cirrhosis, decompensated liver disease, active hepatitis or chronic hepatitis require antiviral treatment.
* 3: A history of immunodeficiency, including HIV positive or other acquired congenital immunodeficiency diseases.
* 4: Chronic renal insufficiency and renal failure.
* 5: Patients who have suffered from or combined with other malignant tumors.
* 6: Myocardial infarction, severe arrhythmia and ≥ grade 2 congestive heart failure (New York Heart Association (NYHA) classification).
* 7: Patients with autoimmune diseases such as systemic lupus erythematosus.
* 8: Complications, need to take drugs with serious liver and kidney damage during treatment, such as tuberculosis.
* 9: Patients who cannot understand the content of the experiment and cannot cooperate and those who refuse to sign the informed consent.
* 10: Those with concomitant diseases or other special circumstances that seriously endanger the safety of patients or affect the completion of the study.
* 11: Combined with neoadjuvant radiotherapy.
* 12: Postoperative follow-up was not completed.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population was patients with locally advanced gastric cancer receiving neoadjuvant chemotherapy.
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-06-28 (Estimated); Study Completion 2024-06-28 (Estimated)

PRIMARY OUTCOMES:
Predictive sensitivity of drug sensitivity | At the end of Cycle 2 (each cycle is 21 days); At the end of Cycle 4 (each cycle is 21 days); Ten days after surgery;
  Consistency ratio between organoid drug screening results and actual clinical observation drug sensitivity.
Predictive specificity of drug sensitivity | At the end of Cycle 2 (each cycle is 21 days); At the end of Cycle 4 (each cycle is 21 days); Ten days after surgery;
  The proportion of inconsistencies between organoid drug screening results and actual clinical observation drug sensitivity.

SECONDARY OUTCOMES:
Concordance between organoids and source tumor tissue | Organoid models were established and compared after passaging 3-5 generations (Three weeks)
  Concordance between organoids and source tumor tissue

CONTACTS AND LOCATIONS:
Overall Officials: Dongbing Zhao, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (1):
- Department of Pancreatic and Gastric Surgical Oncology, National Cancer Center/ National Clinical Research for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College, Beijing, China